CLINICAL TRIAL: NCT06364072
Title: Open-label, Prospective Study to Assess the Safety, Tolerability, Analgesic Effect and Feasibility of Intranasal Sufentanil/Ketamine in Pediatric Patients With Moderate or Severe Pain, in an Acute Care Setting
Brief Title: Safety, Tolerability, Analgesic Effect, and Feasibility of Intranasal CT001 in Pediatric Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cessatech A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDC 01-0202; 2023-504023-63-00 (EU CTIS Number)
Record Dates: First submitted 2024-04-02; First posted 2024-04-15 (Actual); Results first posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT001 (Experimental)
  Interventions: Drug: CT001

INTERVENTIONS:
Drug: CT001 — Intranasal

SUMMARY:
The proposed study aims to investigate the safety, tolerability, analgesic efficacy, and feasibility of intranasal sufentanil/ketamine (CT001) in pediatric participants attending an acute care (i.e. emergency) setting. The study is a part of the clinical development plan for the development of CT001 nasal spray for treatment of acute pain in children.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric participant, age 1 year to 17 years
* Attending an Emergency Department following an injury
* Acute pain of moderate or severe intensity
* Obtained informed consent by parent/guardian and assent from the child if possible and relevant (age dependent)

Exclusion Criteria:

* Participant showing abnormal nasal cavity/airway such as:

  1. major septal deviation
  2. evidence of previous nasal disease or surgery
  3. current significant nasal congestion due to common cold
* Has received treatment with sufentanil and/or ketamine during the last 72 hours
* Known or suspected allergy to ketamine or sufentanil
* Critical, life- or limb-threatening condition requiring immediate management

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 155 (Actual)
Dates: Start 2024-05-27 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Hartshorn, Dr., Principal Investigator — Birmingham Children's Hospital
Locations (7):
- Spain (4):
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Sant Joan de Deu, Barcelona
  - Universidad Autonoma de Madrid (UAM) - Hospital Universitario La Paz (HULP) -, Madrid
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela
- United Kingdom (3):
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham
  - Royal London Hospital, London
  - Sheffield Children's Hospital, Sheffield

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total number of participants enrolled in the study: 155 (83 in Spain and 72 in the United Kingdom).
  There was no screen failures reported, only 1 participant was withdrawn from the study by the investigator due to pending surgical procedures which meant that the patient could not continue on the study.
  There were 155 participants in the full analysis set and in the safety population and 152 participants included in the efficacy analysis.
Groups:
- CT001: All participants received one or potentially two consecutive doses of CT001.
Period: Overall Study
Arm/Group | CT001
Started | 155
Completed | 154
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | CT001
Number analyzed (Participants) | 155
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 68
  Not Hispanic or Latino | 84
  Unknown or Not Reported | 3
Age, Customized [Count of Participants; unit: Participants]
  Age: 1 - < 5 years | 22
  Age: 5 - < 9 years | 38
  Age: 9 - < 18 years | 95
Baseline pain intensity score [Median (Inter-Quartile Range); unit: Score on a scale (0-10)] — Pain intensity was assessed with age-appropriate validated scales. Ages ≥1-<5years: FLACC (Face, Legs, Activity, Cry, Consolability), total score 0-10 (0=no pain, 10=severe pain). Ages ≥5-<9years: Wong-Baker FACES, categories 0,2,4,6,8,10 (range 0-10; higher=worse pain). Ages ≥9years: Numerical Rating Scale (NRS) 0-10 (0=no pain, 10=worst pain imaginable).
  Score on a scale (0-10) | 8 [7 to 9]

OUTCOME MEASURES:

1. Primary Outcome: Sedation
Description: Sedation was assessed by sedation score on the University of Michigan Sedation Scale (UMSS). Scores range from 0 to 4, where 0 = awake/alert, 1 = minimally sedated (tired/sleepy, appropriate response to verbal conversation and/or sound), 2 = moderately sedated (somnolent/sleeping, easily aroused with light tactile stimulation or simple verbal command), 3 = deeply sedated (deep sleep, arousable only with significant physical stimulation), and 4 = unarousable. Lower scores indicate less sedation; higher scores indicate deeper sedation.
Time Frame: At baseline and 10, 15, 20, 30, 45 and 60 min after first IMP administration. If a second IMP dose was needed, sedation score was performed at the timepoints relative to first IMP administration.
Population: Some participants had missing or non-assessable UMSS scores (e.g., early withdrawal, assessment not performed within the prespecified window, or incomplete data).
Measure: Median (Inter-Quartile Range); unit: UMSS score
Arm/Group | CT001
Number analyzed (Participants) | 155
UMSS score
  Baseline | 0 [0 to 0]
  10 min | 0 [0 to 1]
  15 min | 1 [0 to 1]
  20 min | 1 [0 to 1]
  30 min: number analyzed (Participants) | 154
  30 min | 1 [0 to 1]
  45 min: number analyzed (Participants) | 154
  45 min | 0 [0 to 1]
  60 min: number analyzed (Participants) | 154
  60 min | 0 [0 to 1]

2. Primary Outcome: Respiratory Depression
Description: Respiratory depression assessed by respiratory rate.
Time Frame: At baseline and 10, 15, 20, 25, 30, 35, 45, 60 and 75 min after IMP administration.
Population: The number analyzed differs across rows because pain intensity was assessed using age-appropriate scales, and not all participants had evaluable measurements at each time point. Some participants had missing or non-assessable pain scores (e.g., early withdrawal, assessment not performed within the prespecified window, or incomplete data), so they were excluded from the affected row(s), while remaining in the overall analyzed population.
Measure: Median (Standard Deviation); unit: Respiratory rate (rpm)
Arm/Group | CT001
Number analyzed (Participants) | 155
Respiratory rate (rpm)
  Age 1- <5 years, baseline: number analyzed (Participants) | 22
  Age 1- <5 years, baseline | 26 (6.09)
  Age 1- <5 years, 10 min: number analyzed (Participants) | 22
  Age 1- <5 years, 10 min | 24 (5.67)
  Age 1- <5 years, 15 min: number analyzed (Participants) | 18
  Age 1- <5 years, 15 min | 24 (5.27)
  Age 1- <5 years, 20 min: number analyzed (Participants) | 17
  Age 1- <5 years, 20 min | 23 (3.64)
  Age 1- <5 years, 25 min: number analyzed (Participants) | 5
  Age 1- <5 years, 25 min | 21 (3.44)
  Age 1- <5 years, 30 min: number analyzed (Participants) | 22
  Age 1- <5 years, 30 min | 22 (3.87)
  Age 1- <5 years, 35 min: number analyzed (Participants) | 5
  Age 1- <5 years, 35 min | 20 (4)
  Age 1- <5 years, 45 min: number analyzed (Participants) | 22
  Age 1- <5 years, 45 min | 22 (3.59)
  Age 1- <5 years, 60 min: number analyzed (Participants) | 22
  Age 1- <5 years, 60 min | 23.5 (4.24)
  Age 1- <5 years, 75 min: number analyzed (Participants) | 5
  Age 1- <5 years, 75 min | 24 (3.03)
  Age 5- <9 years, baseline: number analyzed (Participants) | 38
  Age 5- <9 years, baseline | 24 (5.05)
  Age 5- <9 years, 10 min: number analyzed (Participants) | 38
  Age 5- <9 years, 10 min | 22 (4.34)
  Age 5- <9 years, 15 min: number analyzed (Participants) | 32
  Age 5- <9 years, 15 min | 20 (3.82)
  Age 5- <9 years, 20 min: number analyzed (Participants) | 25
  Age 5- <9 years, 20 min | 20 (3.28)
  Age 5- <9 years, 25 min: number analyzed (Participants) | 12
  Age 5- <9 years, 25 min | 21.5 (3.52)
  Age 5- <9 years, 30 min: number analyzed (Participants) | 37
  Age 5- <9 years, 30 min | 21 (3.48)
  Age 5- <9 years, 35 min: number analyzed (Participants) | 12
  Age 5- <9 years, 35 min | 23 (3.26)
  Age 5- <9 years, 45 min: number analyzed (Participants) | 36
  Age 5- <9 years, 45 min | 20 (3.42)
  Age 5- <9 years, 60 min: number analyzed (Participants) | 37
  Age 5- <9 years, 60 min | 21 (3.6)
  Age 5- <9 years, 75 min: number analyzed (Participants) | 12
  Age 5- <9 years, 75 min | 22 (3.87)
  Age 9- <18 years, baseline: number analyzed (Participants) | 95
  Age 9- <18 years, baseline | 20 (4.31)
  Age 9- <18 years, 10 min: number analyzed (Participants) | 95
  Age 9- <18 years, 10 min | 20 (4.09)
  Age 9- <18 years, 15 min: number analyzed (Participants) | 84
  Age 9- <18 years, 15 min | 20 (3.43)
  Age 9- <18 years, 20 min: number analyzed (Participants) | 74
  Age 9- <18 years, 20 min | 19 (3.68)
  Age 9- <18 years, 25 min: number analyzed (Participants) | 21
  Age 9- <18 years, 25 min | 19 (3.33)
  Age 9- <18 years, 30 min: number analyzed (Participants) | 95
  Age 9- <18 years, 30 min | 18 (3.13)
  Age 9- <18 years, 35 min: number analyzed (Participants) | 21
  Age 9- <18 years, 35 min | 16 (2.87)
  Age 9- <18 years, 45 min: number analyzed (Participants) | 95
  Age 9- <18 years, 45 min | 18 (3.06)
  Age 9- <18 years, 60 min: number analyzed (Participants) | 94
  Age 9- <18 years, 60 min | 18 (3.18)
  Age 9- <18 years, 75 min: number analyzed (Participants) | 21
  Age 9- <18 years, 75 min | 17 (2.26)

3. Secondary Outcome: Treatment Satisfaction
Description: Treatment satisfaction as assessed by responses to the question: "How satisfied are you with the study drug that you/your child received? Please think about how it helped their pain, how it was given, any side effects, and how quickly you/your child recovered". Respondents answered using a 5-point Likert scale (very unsatisfied (1), unsatisfied (2), neutral (3), satisfied (4), very satisfied (5)).
Time Frame: Prior to Emergency Department discharge (day of IMP administration)
Measure: Median (Inter-Quartile Range); unit: Treatment satistaction score
Arm/Group | CT001
Number analyzed (Participants) | 155
Treatment satistaction score | 5 [5 to 5]

4. Primary Outcome: Peripheral Oxygen Saturation
Description: Peripheral oxygen saturation assessed by oxygen saturation rate (%)
Time Frame: At baseline and 10, 15, 20, 25, 30, 35, 45, 60 and 75 min after IMP administration.
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: Oxygen saturation rate (%)
Arm/Group | CT001
Number analyzed (Participants) | 155
Oxygen saturation rate (%)
  Age 1- <5 years, baseline: number analyzed (Participants) | 22
  Age 1- <5 years, baseline | 98 (1.05)
  Age 1- <5 years, 10 min: number analyzed (Participants) | 22
  Age 1- <5 years, 10 min | 98 (1.15)
  Age 1- <5 years, 15 min: number analyzed (Participants) | 18
  Age 1- <5 years, 15 min | 98 (1.17)
  Age 1- <5 years, 20 min: number analyzed (Participants) | 17
  Age 1- <5 years, 20 min | 98 (1.22)
  Age 1- <5 years, 25 min: number analyzed (Participants) | 5
  Age 1- <5 years, 25 min | 97 (1)
  Age 1- <5 years, 30 min: number analyzed (Participants) | 22
  Age 1- <5 years, 30 min | 98 (1.4)
  Age 1- <5 years, 35 min: number analyzed (Participants) | 5
  Age 1- <5 years, 35 min | 98 (0.89)
  Age 1- <5 years, 45 min: number analyzed (Participants) | 22
  Age 1- <5 years, 45 min | 99 (1.4)
  Age 1- <5 years, 60 min: number analyzed (Participants) | 22
  Age 1- <5 years, 60 min | 98 (1.39)
  Age 1- <5 years, 75 min: number analyzed (Participants) | 5
  Age 1- <5 years, 75 min | 98 (1.64)
  Age 5- <9 years, baseline: number analyzed (Participants) | 38
  Age 5- <9 years, baseline | 98 (1.32)
  Age 5- <9 years, 10 min: number analyzed (Participants) | 38
  Age 5- <9 years, 10 min | 98 (1.5)
  Age 5- <9 years, 15 min: number analyzed (Participants) | 32
  Age 5- <9 years, 15 min | 98 (1.42)
  Age 5- <9 years, 20 min: number analyzed (Participants) | 25
  Age 5- <9 years, 20 min | 98 (1.28)
  Age 5- <9 years, 25 min: number analyzed (Participants) | 12
  Age 5- <9 years, 25 min | 97.5 (1.73)
  Age 5- <9 years, 30 min: number analyzed (Participants) | 37
  Age 5- <9 years, 30 min | 98 (1.44)
  Age 5- <9 years, 35 min: number analyzed (Participants) | 12
  Age 5- <9 years, 35 min | 97 (1.68)
  Age 5- <9 years, 45 min: number analyzed (Participants) | 36
  Age 5- <9 years, 45 min | 98 (1.43)
  Age 5- <9 years, 60 min: number analyzed (Participants) | 37
  Age 5- <9 years, 60 min | 98 (2.08)
  Age 5- <9 years, 75 min: number analyzed (Participants) | 12
  Age 5- <9 years, 75 min | 98.5 (1.9)
  Age 9- <18 years, baseline: number analyzed (Participants) | 95
  Age 9- <18 years, baseline | 99 (1.35)
  Age 9- <18 years, 10 min: number analyzed (Participants) | 94
  Age 9- <18 years, 10 min | 99 (1.54)
  Age 9- <18 years, 15 min: number analyzed (Participants) | 84
  Age 9- <18 years, 15 min | 98 (1.52)
  Age 9- <18 years, 20 min: number analyzed (Participants) | 74
  Age 9- <18 years, 20 min | 98 (1.55)
  Age 9- <18 years, 25 min: number analyzed (Participants) | 21
  Age 9- <18 years, 25 min | 98 (1.5)
  Age 9- <18 years, 30 min: number analyzed (Participants) | 95
  Age 9- <18 years, 30 min | 98 (1.61)
  Age 9- <18 years, 35 min: number analyzed (Participants) | 21
  Age 9- <18 years, 35 min | 98 (1.46)
  Age 9- <18 years, 45 min: number analyzed (Participants) | 95
  Age 9- <18 years, 45 min | 98 (2.07)
  Age 9- <18 years, 60 min: number analyzed (Participants) | 94
  Age 9- <18 years, 60 min | 98 (2.22)
  Age 9- <18 years, 75 min: number analyzed (Participants) | 21
  Age 9- <18 years, 75 min | 98 (2.23)

5. Primary Outcome: Cardiovascular Stability
Description: Cardiovascular stability assessed by pulse rate (bpm)
Time Frame: At baseline and 10, 15, 20, 25, 30, 35, 45, 60 and 75 min after IMP administration.
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: Beats per minute
Arm/Group | CT001
Number analyzed (Participants) | 155
Beats per minute
  Age 1- <5 years, baseline: number analyzed (Participants) | 22
  Age 1- <5 years, baseline | 117 (22.69)
  Age 1- <5 years, 10 min: number analyzed (Participants) | 22
  Age 1- <5 years, 10 min | 108 (17.78)
  Age 1- <5 years, 15 min: number analyzed (Participants) | 18
  Age 1- <5 years, 15 min | 111 (18.37)
  Age 1- <5 years, 20 min: number analyzed (Participants) | 17
  Age 1- <5 years, 20 min | 109 (16.7)
  Age 1- <5 years, 25 min: number analyzed (Participants) | 5
  Age 1- <5 years, 25 min | 118 (9.84)
  Age 1- <5 years, 30 min: number analyzed (Participants) | 22
  Age 1- <5 years, 30 min | 109 (16.5)
  Age 1- <5 years, 35 min: number analyzed (Participants) | 5
  Age 1- <5 years, 35 min | 117 (7.95)
  Age 1- <5 years, 45 min: number analyzed (Participants) | 22
  Age 1- <5 years, 45 min | 110 (12.91)
  Age 1- <5 years, 60 min: number analyzed (Participants) | 22
  Age 1- <5 years, 60 min | 109 (12.73)
  Age 1- <5 years, 75 min: number analyzed (Participants) | 5
  Age 1- <5 years, 75 min | 110 (9.56)
  Age 5- <9 years, baseline: number analyzed (Participants) | 38
  Age 5- <9 years, baseline | 103.5 (14.92)
  Age 5- <9 years, 10 min: number analyzed (Participants) | 38
  Age 5- <9 years, 10 min | 97.5 (11.74)
  Age 5- <9 years, 15 min: number analyzed (Participants) | 32
  Age 5- <9 years, 15 min | 96.5 (13.88)
  Age 5- <9 years, 20 min: number analyzed (Participants) | 25
  Age 5- <9 years, 20 min | 93 (12.75)
  Age 5- <9 years, 25 min: number analyzed (Participants) | 12
  Age 5- <9 years, 25 min | 96.5 (12.59)
  Age 5- <9 years, 30 min: number analyzed (Participants) | 37
  Age 5- <9 years, 30 min | 95 (14.48)
  Age 5- <9 years, 35 min: number analyzed (Participants) | 12
  Age 5- <9 years, 35 min | 93.5 (15.34)
  Age 5- <9 years, 45 min: number analyzed (Participants) | 36
  Age 5- <9 years, 45 min | 91 (13.97)
  Age 5- <9 years, 60 min: number analyzed (Participants) | 37
  Age 5- <9 years, 60 min | 92 (13.07)
  Age 5- <9 years, 75 min: number analyzed (Participants) | 12
  Age 5- <9 years, 75 min | 105 (14.43)
  Age 9- <18 years, baseline: number analyzed (Participants) | 95
  Age 9- <18 years, baseline | 90 (15.02)
  Age 9- <18 years, 10 min: number analyzed (Participants) | 95
  Age 9- <18 years, 10 min | 87 (15.71)
  Age 9- <18 years, 15 min: number analyzed (Participants) | 84
  Age 9- <18 years, 15 min | 85 (13.6)
  Age 9- <18 years, 20 min: number analyzed (Participants) | 74
  Age 9- <18 years, 20 min | 83 (15.17)
  Age 9- <18 years, 25 min: number analyzed (Participants) | 21
  Age 9- <18 years, 25 min | 86 (13.49)
  Age 9- <18 years, 30 min: number analyzed (Participants) | 95
  Age 9- <18 years, 30 min | 80 (15.09)
  Age 9- <18 years, 35 min: number analyzed (Participants) | 21
  Age 9- <18 years, 35 min | 83 (14.46)
  Age 9- <18 years, 45 min: number analyzed (Participants) | 95
  Age 9- <18 years, 45 min | 83 (15.11)
  Age 9- <18 years, 60 min: number analyzed (Participants) | 94
  Age 9- <18 years, 60 min | 82 (14.77)
  Age 9- <18 years, 75 min: number analyzed (Participants) | 21
  Age 9- <18 years, 75 min | 80 (14.36)

6. Primary Outcome: Number of Reported Adverse Events
Description: Number of reported adverse events.
Time Frame: Through study completion; up to 7 days
Measure: Number; unit: Adverse events
Arm/Group | CT001
Number analyzed (Participants) | 155
Adverse events | 132

7. Primary Outcome: Number of Adverse Events (AEs) Reported Per Participant
Description: Number of adverse events (AEs) reported per participant.
Time Frame: Through study completion; up to 7 days
Measure: Number; unit: Adverse event per participant
Arm/Group | CT001
Number analyzed (Participants) | 155
Adverse event per participant | 0.85

8. Secondary Outcome: Feasibility (Acceptance of Nasal Administration)
Description: Feasibility (i.e. acceptance of nasal administration) was addressed by the healthcare staff asking the participant: "If you were in this situation again and needed pain medication, would you like to receive the nasal spray (relative to an injection, tablet or suppository for the pain)?' If not possible by the participant, the parent/legal guardian assessed nasal acceptability. Answers were "yes, "no", "I don't know".
Time Frame: Prior to Emergency Department discharge (day of IMP administration)
Measure: Count of Participants; unit: Participants
Arm/Group | CT001
Number analyzed (Participants) | 153
Participants
  "Yes" | 143
  "No" | 4
  "I don't know" | 6

9. Secondary Outcome: Medication Errors
Description: Medication errors, defined as any deviation in the IMP administration instructions that resulted in higher or lower dose than planned. Examples may include erroneous priming of the pump, too few/many pumps administered, etc.
Time Frame: Assessed immediately post IMP administration
Measure: Number; unit: Participants
Arm/Group | CT001
Number analyzed (Participants) | 155
Participants
  Reported number of participants with medication errors | 3
  Number of participants with no medication errors | 152

10. Secondary Outcome: Maximum Change From Baseline in Pain Intensity Within 30 Min Post (First) IMP Administration.
Description: Pain intensity was assessed with age-appropriate validated scales. Ages ≥1-<5years: FLACC (Face, Legs, Activity, Cry, Consolability), total score 0-10 (0=no pain, 10=severe pain). Ages ≥5-<9years: Wong-Baker FACES, categories 0,2,4,6,8,10 (range 0-10; higher=worse pain). Ages ≥9years: Numerical Rating Scale (NRS) 0-10 (0=no pain, 10=worst pain imaginable).
Time Frame: 30 min post (first) IMP administration
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | CT001
Number analyzed (Participants) | 152
Scores on a scale | -6 [-8 to -4]

11. Secondary Outcome: Number of Participants That Achieved a 30% (or More) Reduction in Pain Intensity Relative to Baseline
Description: as for outcome 10
Time Frame: within 30 min post (first) IMP administration.
Measure: Count of Participants; unit: Participants
Arm/Group | CT001
Number analyzed (Participants) | 152
Participants | 145

12. Secondary Outcome: Change From Baseline in Pain Intensity
Description: as for outcome 10
Time Frame: at 10, 15, 20, 30, 45 and 60 min post last dose of IMP administration.
Population: Only patients who had evaluable pain-intensity measurements for the relevant endpoint/time point are included in this outcome measure. Although 155 patients were treated and included in the overall safety population, some did not have a valid post-baseline assessment (e.g., missing measurement, assessment outside the prespecified window, early discontinuation, or other clinical/technical reasons).
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | CT001
Number analyzed (Participants) | 152
Scores on a scale
  10 min | -2 [-4 to -1]
  15 min | -4 [-6 to -3]
  20 min (1 dose) | -5 [-7 to -4]
  25 min (2 doses) | -4 [-6 to -3]
  30 min | -6 [-8 to -4]
  35 min (2 doses) | -6 [-8 to -5]
  45 min | -6 [-8 to -5]
  60 min | -6 [-8 to -5]
  75 min (2 doses) | -7 [-8 to -5]

13. Primary Outcome: Local Nasal Irritation
Description: The number of participants with nasal irritation was summarised using counts of participants for each timepoint (30 and 60 min post IMP administration) by type of nasal irritation.
Time Frame: 30 and 60 min post IMP administration
Measure: Number; unit: Number of participants
Arm/Group | CT001
Number analyzed (Participants) | 154
Number of participants
  Itching, 30 min post IMP | 16
  Itching, 60 min post IMP | 7
  Nasal discharge, 30 min post IMP | 0
  Nasal discharge, 60 min post IMP | 1
  Other nasal irritation, 30 min post IMP | 3
  Other nasal irritation, 60 min post IMP | 1
  Redness, 30 min post IMP | 2
  Redness, 60 min post IMP | 1
  Sneezing, 30 min post IMP | 1
  Sneezing, 60 min post IMP | 0

14. Primary Outcome: Analgesic Effect
Description: Number and proportion of participants that respond to the treatment relative to baseline (i.e. reduction in pain score to 4 or below). Pain intensity was assessed with age-appropriate validated scales. Ages ≥1-<5years: FLACC (Face, Legs, Activity, Cry, Consolability), total score 0-10 (0=no pain, 10=severe pain). Ages ≥5-<9years: Wong-Baker FACES, categories 0,2,4,6,8,10 (range 0-10; higher=worse pain). Ages ≥9years: Numerical Rating Scale (NRS) 0-10 (0=no pain, 10=worst pain imaginable).
Time Frame: At baseline and at 15 and 30 min post first IMP dose
Population: As the results include two time points, some participants are represented in more than one category.
Measure: Count of Participants; unit: Participants
Arm/Group | CT001
Number analyzed (Participants) | 152
Participants
  Participants with pain intensity <=4 at 15min post first dose of CT001 | 82
  Participants with pain intensity > 4 at 15min post first dose of CT001 | 70
  Participants with pain intensity <=4 at 30min post first dose of CT001 | 134
  Participants with pain intensity > 4 at 30min post first dose of CT001 | 18

15. Secondary Outcome: Number of Children Receiving Additional Analgesics
Description: Number of children receiving additional analgesics.
Time Frame: During the 60 min period post last dose of IMP
Measure: Number; unit: participants
Arm/Group | CT001
Number analyzed (Participants) | 139
participants | 17

ADVERSE EVENTS:
Time Frame: Through study completion; up to 7 days
Arm/Group | CT001
All-Cause Mortality (participants affected / at risk) | 0/155
Serious Adverse Events (participants affected / at risk) | 4/155
Other Adverse Events (participants affected / at risk) | 73/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CT001 (N=155)
Hospitalisation (Surgical and medical procedures) | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CT001 (N=155)
Lacrimation increased (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 25
Product use complaint (Injury, poisoning and procedural complications) | 19
Decreased appetite (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 22
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Abnormal behaviour (Psychiatric disorders) | 1
Anger (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Euphoric mood (Psychiatric disorders) | 1
Mood altered (Psychiatric disorders) | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 2
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 13
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 4
Erythema (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 10
Hospitalisation (Surgical and medical procedures) | 4
Hot flush (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-18): https://cdn.clinicaltrials.gov/large-docs/72/NCT06364072/Prot_SAP_000.pdf